CLINICAL TRIAL: NCT05718297
Title: A Multicentre, Randomised, Phase II Trial of Brigatinib Consolidation Versus Observation or Durvalumab in Patients with Unresectable Stage III NSCLC and ALK-rearrangement, After Definitive Chemo-radiotherapy
Brief Title: Brigatinib Post Definitive Chemo-radiotherapy in Patients with ALK-fusion Non-small Cell Lung Cancer
Acronym: BOUNCE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Despite our efforts, the trial faced challenges like a longer activation period and slower accrual. We proposed a redesign, but TAKEDA withdrew. As a non-profit organisation, we can't continue without TAKEDA's support and must discontinue the trial.
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 21-21
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: NSCLC, Stage III; ALK-rearrangement
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — brigatinib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): Brigatinib 180 mg once daily p.o., with seven day lead-in at 90 mg once daily, for 3 years or until progression of disease, or unacceptable toxicities or withdrawal of consent
  Interventions: Drug: Brigatinib
- Control arm (Active Comparator): Patients in the control arm will be observational, or, as per investigators choice, patients may receive durvalumab, administered within the label in the respective country.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Brigatinib — Brigatinib is administered for 3 years or until progression of disease, or unacceptable toxicities or withdrawal of consent, whatever occurs first. After the treatment period of 3 years, patient's ongoing treatment will be managed according to local standard and best clinical practice.
  Brigatinib should be taken approximately at the same time each day. It may be taken with or without food. Patients shall be instructed to swallow the tablets whole and not crush or chew them.
  Arms: Experimental arm
Drug: Durvalumab — Patients in the control arm will be observational, or, as per investigators choice, patients may receive durvalumab, administered within the label in the respective country.
  Arms: Control arm

SUMMARY:
BOUNCE is an international multicentre randomised phase II trial. The trial treatment consists of brigatinib 180 mg once daily p.o., with seven day lead-in at 90 mg once daily, for 3 years or until progression of disease. The primary objective of this trial is to evaluate the efficacy in terms of progression-free survival (PFS) for brigatinib consolidation, compared to observation/durvalumab, in patients with unresectable stage III NSCLC and ALK-rearrangement who completed definitive chemo-radiotherapy without disease progression.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for enrolment

* Pathologically documented, treatment naïve unresectable stage III NSCLC
* Documented ALK-fusion, tested locally on tumour tissue by a validated method (DNA NGS, RNA NGS, FISH, IHC, or ctDNA)
* ECOG Performance Status 0-1
* Age ≥18 years
* Patient is a candidate to receive chemo-radiotherapy, as per investigator's assessment (including adequate haematological, renal and liver function as per local guidelines).
* Women of childbearing potential, including women who had their last menstruation in the last 2 years, must have a negative urinary or serum pregnancy test within 5 weeks before enrolment.
* Ability to comply with the trial protocol, in the investigator's judgment.
* Written IC for trial participation must be signed and dated by the patient and the investigator prior to any trial-related intervention, including the submission of mandatory biomaterial.

Eligibility criteria for randomisation Randomisation of eligible patients must occur within 8 weeks after the last radiotherapy fraction.

* Completion of thoracic radiotherapy
* Non-PD at restaging
* Adequate haematological function
* Adequate renal function
* Adequate liver and pancreatic function
* Women of childbearing potential, including women who had their last menstruation in the last 2 years, must have a negative urinary or serum pregnancy test before randomisation and should be repeated within 3 days before the first dose of brigatinib.
* No radiation-pneumonitis of grade ≥2
* All other AEs from previous chemo-radiotherapy resolved to grade <2 (except for alopecia)
* ECOG 0-2
* No major surgery as defined by the investigator within 4 weeks of the the first planned dose of brigatinib.

Minor surgical procedures such as catheter placement or minimally invasive biopsies are allowed.

* No systemic treatment with strong cytochrome p-450 (cyp)3a inhibitors, strong cyp3a inducers, or moderate cyp3a inducers within 14 days before randomisation.

Exclusion Criteria:

* Diagnosis of another primary malignancy other than NSCLC. With the exception of adequately treated non-melanoma skin cancer or cervical cancer in situ; definitively treated non-metastatic prostate cancer; or patients with another primary malignancy who are definitively relapse-free with at least 3 years since the diagnosis of the other primary malignancy.
* Prior treatment for NSCLC
* Any evidence of stage IV NSCLC
* Significant, uncontrolled, or active cardiovascular disease
* Uncontrolled hypertension Patients with hypertension should be under treatment on study entry to control blood pressure.
* History or the presence at baseline of pulmonary interstitial disease, drug-related pneumonitis.
* Ongoing or active infection, including, but not limited to, the requirement for intravenous antibiotics.
* Malabsorption syndrome or other GI illness that could affect oral absorption of brigatinib.
* Known or suspected hypersensitivity to brigatinib or its excipients.
* Any concurrent medical condition which, in the opinion of the investigator, would compromise patient safety or interfere with the evaluation of brigatinib.
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
* Women who are pregnant or in the period of lactation.
* Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the trial until at least 4 months after the last dose of protocol treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival, according to RECIST v1.1, evaluated in the ITT cohort. PFS will be compared between the two arms. | From the date of enrolment until last tumour assessment (approximately 45-48 months after enrolment of the first patient)
  defined as the time from the date of randomisation until documented progression (according to RECIST v1.1) or death, if progression is not documented

SECONDARY OUTCOMES:
Overall survival | From the date of enrolment until last tumour assessment (approximately 45-48 months after enrolment of the first patient)
  Defined as the time from the date of randomisation until death from any cause
CNS-relapse-free survival | From the date of enrolment until last tumour assessment (approximately 45-48 months after enrolment of the first patient)
  Defined as the time from the date of randomisation until documented CNS-relapse, at the first disease progression, according to RECIST v1.1 or death from any cause, if CNS-relapse is not documented
Patterns of disease progression | From the date of enrolment until last tumour assessment (approximately 45-48 months after enrolment of the first patient)
  Defined as the site of first progression after randomisation: None, locoregional, distant (bone, brain, liver, etc.) or both locoregional and distant.
Toxicity according to CTCAE v5.0 | From the date of enrolment until last tumour assessment (approximately 45-48 months after enrolment of the first patient)
  All safety parameters from enrolment will be summarised in tables to evaluate the toxicity/safety profile of the protocol treatment based on:
  * Adverse events according to CTCAE v5.0 (any-cause as well as treatment-related) including adverse events leading to dose interruptions, withdrawal of protocol treatment, and death
  * Severe, serious, and selected adverse events
  * Deaths
  * Laboratory parameters and abnormalities, and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Rafal Dziadziuszko, MD, Study Chair — Dept. of Oncology and Radiotherapy, Medical University of Gdansk
Locations (20):
- France (3):
  - CHU Angers, Angers
  - Caen - CHU, Caen
  - Hôpital de Marseille, Marseille
- Italy (7):
  - IRCCS Instituto Tumori Giovanni Paolo II, Bari
  - IRCCS - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola
  - AOU Maggiore della Carità, Novara
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Santa Maria della Misericordia Hospital, Perugia
  - AULSS2 Marca Trevigiana Treviso, Treviso
  - Universita di Verona - Department of Medicine, Verona
- Medical University Gdansk, Gdansk, Poland
- Spain (7):
  - Hospital Universitario Dr Balmis Alicante - ISABIAL, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Basurto, Bilbao
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Universitario Lucus Augusti, Lugo
  - H. Puerta de Hierro Majadahonda, Majadahonda
- United Kingdom (2):
  - Royal Marsden Hospital (Fulham Road), London
  - Royal Marsden Hospital (Sutton), London

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP